CLINICAL TRIAL: NCT06910202
Title: Effects of Cigarette and E-cigarette Flavors on Substitutability in the Experimental Tobacco Marketplace (20-008)
Brief Title: Effects of Cigarette and E-cigarette Flavors on Substitutability in the ETM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VT IRB #25-185; 5P01CA200512-09 (NIH)
Record Dates: First submitted 2025-03-07; First posted 2025-04-04 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-02

CONDITIONS: Cigarette Smoking Behavior
Keywords: Cigarettes; E-cigarettes; Experimental Tobacco Marketplace; Substitutability; Flavors
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Menthol cigarette smokers (Experimental): Menthol cigarette smokers will complete questionnaires on a computer, sample a range of tobacco products, and purchase tobacco products in an online store under four different scenarios: a) cigarette flavor restricted and e-cigarette flavor restricted, b) cigarette flavor unrestricted and e-cigarette flavor restricted, c) cigarette flavor restricted and e-cigarette flavor unrestricted, d) cigarette flavor unrestricted and e-cigarette flavor unrestricted.
  Interventions: Behavioral: Manipulation of nicotine/tobacco product price and availability

INTERVENTIONS:
Behavioral: Manipulation of nicotine/tobacco product price and availability — This study does involve experimental manipulation of nicotine/tobacco product price and availability to understand consumers' behavior. Participants will be provided with a commercially available e-cigarette to use during the study, if they wish.
  Every participant will purchase tobacco products in an online store under four different scenarios: a) cigarette flavor restricted and e-cigarette flavor restricted, b) cigarette flavor unrestricted and e-cigarette flavor restricted, c) cigarette flavor restricted and e-cigarette flavor unrestricted, d) cigarette flavor unrestricted and e-cigarette flavor unrestricted.

SUMMARY:
In 2009, the FDA banned all flavored conventional cigarettes except menthol. While no such ban exists for e-cigarettes, proposals have emerged in several regions. Flavors are key targets for tobacco control policy, making it crucial to understand their role in substitution.The first wave of the PATH study found that 80% of youth, 73% of young adults, and 29% of older smokers used flavored products. Over 80% of young adults first used flavored tobacco, compared to about 50% of adults. Among ever-users, current tobacco use was 32% higher if their first product was flavored.One study reported that 75% of flavored product users would quit if flavors were removed. These findings highlight the importance of user type in shaping policy and raise the question of whether banning flavors would increase quitting or drive substitution.

The Experimental Tobacco Marketplace (ETM) is a novel method for estimating the effects of new tobacco policies and products on consumption and substitution. By experimentally controlling product mix, prices, and policies, ETM simulates "real-world" conditions to assess potential policy impacts.This methodology has been used to study various policies in adult smokers under this grant: nicotine dose variations (Study 1), tobacco taxes and subsidies (Study 2), and workplace restrictions (Study 3). Study 1 found that cigarette and e-cigarette substitutability increased with e-liquid nicotine strength, with 24mg/mL showing the highest substitution. Study 2 showed that cigarette taxes reduced cigarette purchases and increased e-liquid purchases, while e-liquid subsidies increased e-liquid purchases but did not affect cigarette consumption.

No study to date has experimentally examined the effects of flavored tobacco products availability on consumer behavior. The rationale for this specific proposal is to explore prospectively the possible consequences of a flavor ban on consumption and substitution with tobacco products. The results might inform tobacco control policies.

DETAILED DESCRIPTION:
This study does not involve any smoking cessation interventions. This study does involve experimental manipulation of nicotine/tobacco product price and availability to understand consumers' behavior. Participants will be provided with a commercially available e-cigarette to use during the study, if they wish.

This study uses a within subject design. Menthol cigarette smokers will complete questionnaires on a computer, sample a range of tobacco products, and purchase tobacco products in an online store under four different scenarios: a) cigarette flavor restricted and e-cigarette flavor restricted, b) cigarette flavor unrestricted and e-cigarette flavor restricted, c) cigarette flavor restricted and e-cigarette flavor unrestricted, d) cigarette flavor unrestricted and e-cigarette flavor unrestricted.

Participants will complete a 1) consent and assessment session, and a product sampling phase, 2) an ETM session and a 3) follow-up session:

In the consent and initial assessment session, participants will go through standard consent procedures and then provide a breath sample to confirm recent levels of smoking. They may be asked to provide a urine sample for an analysis of cotinine content. Participants will complete a timeline follow back to assess previous month's recent smoking, e-cigarette use, and consumption of nicotine products, and to determine the ETM budget. A Qualtrics survey will administer demographics questions, smoking assessments (Questionnaire on Smoking Urges-Brief, Minnesota Nicotine Withdrawal Scale, Fagerstrom Test of Nicotine Dependence, Perceived Health Risk for cigarettes and e-cigarettes), and delay discounting tasks. At the end of the session, participants will experience a trial of the ETM that will be used in the next session.

For the 7-day sampling phase, they will be provided a list of available flavors and identify 5 that they would like to try. They will leave with a sample of each of the 5 flavors to try during the next few days. Participants will also be provided with a sample of any other tobacco product they wish to examine and try. They may sample any products in the smoking lab before they leave.

In the ETM session, participants will buy tobacco products to use throughout the next 7 days. Participants will complete a total of 40 purchasing trials each for 7 days' worth of products. They will be exposed to 4 conditions with all cigarettes increasing in price and repeat the same conditions with all e-liquids increasing in price across trials. A balanced Latin square design will be used to present the following conditions:

In the Cigarette Flavor Restricted, only conventional tobacco cigarettes will be available. In the Cigarette Flavor Unrestricted, tobacco and menthol cigarettes will be available. In the E-Cigarette Flavor Restricted, only tobacco flavor e-liquids will be available. In the E- Cigarette Flavor Unrestricted, tobacco flavor e-liquid and a variety of other flavors will be available from five broad categories: tobacco, fruit, dessert, menthol, and coffee. A range of other tobacco products will be available across conditions, such as snus, lozenge, gums, dip, and nicotine pouch.

3) In the follow-up session, participants will be able to return the e-cigarette if they wish. They will answer Perceived Health Risk assessments, complete hypothetical purchase tasks for cigarettes and e-cigarettes, rank order the products they sampled, and complete a liking scale for every tobacco product.

We will summarize demographic characteristics (e.g., age, race, income) and smoking-related measures (e.g., FTCD, QSU, PHR) using means, standard deviations, and percentages. For each product category in the ETM, we will test whether policy restrictions differentially influence purchasing of cigarettes, e-cigarettes, oral tobacco/nicotine products, and NRT products.

We will use hierarchical linear regression to evaluate differences in purchasing behavior, including a three-way interaction among the cigarette policy condition, the e-cigarette policy condition, and the log-transformed manipulated commodity price, with random intercepts for individuals. Model selection will be performed to identify the best-supported combination of predictors and interaction terms. We will conduct an exhaustive model search and select the optimal model based on the lowest Bayesian Information Criterion (BIC). Model posterior probabilities will be calculated using BIC following Barbieri and Berger [29].

Model summary statistics will be reported using Type III sums of squares and Kenward-Roger degrees of freedom [30]. All analyses will be performed in R (Version 4.3.0) [31], and statistical significance will be defined as p < 0.05.

Additional analyses may be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Be between 21 and 65 years of age
* Cigarette smokers

  * Smoke cigarettes daily (≥ 5 cigarettes/day)
  * Do not use e-cigarettes regularly (no more than 9 times in the last month)
  * Be willing to try e-cigarettes

Exclusion Criteria:

* Pregnant or lactating women
* Plans to move out of the area
* Use of prescription medication that might affect smoking or nicotine metabolism
* Unmanaged medical or psychiatric conditions
* Plans to quit smoking within the next 30 days
* This study will focus on cigarette smokers and dual users. We will not include individuals under the age of 21 in compliance with Virginia state law. Minors, pregnant women, prisoners, and adults not capable to consent on their own behalf will be excluded from this study.

  1. Minors, as defined by state law where the study is performed (infants, children, teenagers)
  2. Pregnant women (can be included in minimal risk studies by mentioning in section 13.1)
  3. Prisoners (including all incarcerated individuals)
  4. Adults not capable to consent on their own behalf

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas Lemos, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pope DA, Poe L, Stein JS, Kaplan BA, DeHart WB, Mellis AM, Heckman BW, Epstein LH, Chaloupka FJ, Bickel WK. The Experimental Tobacco Marketplace: Demand and Substitutability as a Function of Cigarette Taxes and e-Liquid Subsidies. Nicotine Tob Res. 2020 Apr 21;22(5):782-790. doi: 10.1093/ntr/ntz116. PMID 31350894
- [Background] Pope DA, Poe L, Stein JS, Kaplan BA, Heckman BW, Epstein LH, Bickel WK. Experimental tobacco marketplace: substitutability of e-cigarette liquid for cigarettes as a function of nicotine strength. Tob Control. 2019 Mar;28(2):206-211. doi: 10.1136/tobaccocontrol-2017-054024. Epub 2018 Apr 18. PMID 29669748
- [Background] Bickel WK, Pope DA, Kaplan BA, DeHart WB, Koffarnus MN, Stein JS. Electronic cigarette substitution in the experimental tobacco marketplace: A review. Prev Med. 2018 Dec;117:98-106. doi: 10.1016/j.ypmed.2018.04.026. Epub 2018 Apr 24. PMID 29702131
- [Background] Harrell MB, Loukas A, Jackson CD, Marti CN, Perry CL. Flavored Tobacco Product Use among Youth and Young Adults: What if Flavors Didn't Exist? Tob Regul Sci. 2017 Apr;3(2):168-173. doi: 10.18001/TRS.3.2.4. PMID 28775996
- [Background] Villanti AC, Johnson AL, Ambrose BK, Cummings KM, Stanton CA, Rose SW, Feirman SP, Tworek C, Glasser AM, Pearson JL, Cohn AM, Conway KP, Niaura RS, Bansal-Travers M, Hyland A. Flavored Tobacco Product Use in Youth and Adults: Findings From the First Wave of the PATH Study (2013-2014). Am J Prev Med. 2017 Aug;53(2):139-151. doi: 10.1016/j.amepre.2017.01.026. Epub 2017 Mar 16. PMID 28318902
- [Background] Providenceri.com. Providence Tobacco Laws Go Into Effect January 3. Healthy Communities 2013. https://www.providenceri.com/healthy-communities/providence-tobacco-laws-go-into-effect-january-3.
- [Background] FOX32News. Illinois attorney general: ban e-cigarette flavors. 2014. http://www.myfoxchicago.com/story/26238470/illinois-attorney-general-ban-e-cigarette-flavors. Accessed 11-3-14.
- [Background] Durkin E. Bill would ban sale of flavored e-cigarettes. Celeste Katz Daily Politics. New York: New York Daily News; 2014.

RESULTS

PARTICIPANT FLOW:
Groups:
- Menthol Cigarette Smokers: Menthol cigarette smokers will complete questionnaires on a computer, sample a range of tobacco products, and purchase tobacco products in an online store under four different scenarios: a) cigarette flavor restricted and e-cigarette flavor restricted, b) cigarette flavor unrestricted and e-cigarette flavor restricted, c) cigarette flavor restricted and e-cigarette flavor unrestricted, d) cigarette flavor unrestricted and e-cigarette flavor unrestricted.
  Manipulation of nicotine/tobacco product price and availability: This study does involve experimental manipulation of nicotine/tobacco product price and availability to understand consumers' behavior. Participants will be provided with a commercially available e-cigarette to use during the study, if they wish.
  Every participant will purchase tobacco products in an online store under four different scenarios: a) cigarette flavor restricted and e-cigarette flavor restricted, b) cigarette flavor unrestricted and e-cigarette flavor restricted, c) cigarette flavor restricted and e-cigarette flavor unrestricted, d) cigarette flavor unrestricted and e-cigarette flavor unrestricted.
Period: Overall Study
Arm/Group | Menthol Cigarette Smokers
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Menthol Cigarette Smokers
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Nicotine/Tobacco Products Substitution
Description: The outcome measure of substitution will be collected and modeled using a virtual store. Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price (cigarette type depending on condition). Other product prices will remain at market price. Substitutability occurs as a function of different flavor conditions. The degree to which other nicotine/tobacco products substitute for usual cigarettes under varying price and flavor restriction conditions will be assessed. Mixed-effects hierarchical linear regression will be used to evaluate purchasing behavior. The model includes a three-way interaction (cigarette policy × e-cigarette policy × log(price)) and a random effect for participant. Model selection based on Bayesian Information Criterion (BIC).
Time Frame: During the intervention, session 2 (1 day per participant)
Population: All participants who completed at least one of the experimental purchase scenarios. Missing data for participants who did not complete a condition are noted in the outcome data table.
Measure: Mean (Standard Error); unit: mg of nicotine purchased
Arm/Group | Menthol Cigarette Smokers
Number analyzed (Participants) | 25
mg of nicotine purchased
  Cig & E-cig flavors restricted; Cig price increased; product: Cigarette: number analyzed (Participants) | 24
  Cig & E-cig flavors restricted; Cig price increased; product: Cigarette | 1326.25 (290.72)
  Cig & E-cig flavors restricted; Cig price increased; product: E-Liquid: number analyzed (Participants) | 24
  Cig & E-cig flavors restricted; Cig price increased; product: E-Liquid | 206 (57.29)
  Cig & E-cig flavors restricted; Cig price increased; product: NRT: number analyzed (Participants) | 24
  Cig & E-cig flavors restricted; Cig price increased; product: NRT | 120.83 (39.18)
  Cig & E-cig flavors restricted; Cig price increased; product: OTNP: number analyzed (Participants) | 24
  Cig & E-cig flavors restricted; Cig price increased; product: OTNP | 46.79 (26.20)
  Cig & E-cig flavors unrestricted; Cig price increased; product: Cigarette | 2177.2 (330.38)
  Cig & E-cig flavors unrestricted; Cig price increased; product: E-Liquid | 528 (150.78)
  Cig & E-cig flavors unrestricted; Cig price increased; product: NRT | 41.28 (16.49)
  Cig & E-cig flavors unrestricted; Cig price increased; product: OTNP | 20.72 (12.57)
  Cig flavor restricted, E-cig flavor unrestricted; Cig price increased; product: Cigarette | 1373.2 (316.93)
  Cig flavor restricted, E-cig flavor unrestricted; Cig price increased; product: E-Liquid | 921.6 (277.03)
  Cig flavor restricted, E-cig flavor unrestricted; Cig price increased; product: NRT | 74.72 (28.75)
  Cig flavor restricted, E-cig flavor unrestricted; Cig price increased; product: OTNP | 16.16 (7.55)
  Cig flavor unrestricted, E-cig flavor restricted; Cig price increased; product: Cigarette | 2182 (307.20)
  Cig flavor unrestricted, E-cig flavor restricted; Cig price increased; product: E-Liquid | 126.72 (40.22)
  Cig flavor unrestricted, E-cig flavor restricted; Cig price increased; product: NRT | 96.8 (48.93)
  Cig flavor unrestricted, E-cig flavor restricted; Cig price increased; product: OTNP | 19.08 (9.34)
  Cig & E-cig flavors restricted; E-cig price increased; product: Cigarette | 1590 (332.35)
  Cig & E-cig flavors restricted; E-cig price increased; product: E-Liquid | 164.16 (44.74)
  Cig & E-cig flavors restricted; E-cig price increased; product: NRT | 121.44 (53.82)
  Cig & E-cig flavors restricted; E-cig price increased; product: OTNP | 50.76 (35.23)
  Cig & E-cig flavors unrestricted; E-cig price increased; product: Cigarette: number analyzed (Participants) | 24
  Cig & E-cig flavors unrestricted; E-cig price increased; product: Cigarette | 2674.58 (503.29)
  Cig & E-cig flavors unrestricted; E-cig price increased; product: E-Liquid: number analyzed (Participants) | 24
  Cig & E-cig flavors unrestricted; E-cig price increased; product: E-Liquid | 327 (103.98)
  Cig & E-cig flavors unrestricted; E-cig price increased; product: NRT: number analyzed (Participants) | 24
  Cig & E-cig flavors unrestricted; E-cig price increased; product: NRT | 37.17 (16.01)
  Cig & E-cig flavors unrestricted; E-cig price increased; product: OTNP: number analyzed (Participants) | 24
  Cig & E-cig flavors unrestricted; E-cig price increased; product: OTNP | 9.33 (5.16)
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: Cigarette: number analyzed (Participants) | 24
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: Cigarette | 1774.17 (425.03)
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: E-Liquid: number analyzed (Participants) | 24
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: E-Liquid | 821 (248.81)
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: NRT: number analyzed (Participants) | 24
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: NRT | 58 (24.64)
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: OTNP: number analyzed (Participants) | 24
  Cig flavor restricted, E-cig flavor unrestricted; E-cig price increased; product: OTNP | 14.21 (7.53)
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: Cigarette: number analyzed (Participants) | 24
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: Cigarette | 3312.92 (491.67)
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: E-Liquid: number analyzed (Participants) | 24
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: E-Liquid | 116 (37.08)
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: NRT: number analyzed (Participants) | 24
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: NRT | 62.33 (22.86)
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: OTNP: number analyzed (Participants) | 24
  Cig flavor unrestricted, E-cig flavor restricted; E-cig price increased; product: OTNP | 13.42 (7.39)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Menthol Cigarette Smokers
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
This project is a secondary analysis of data originally collected under IRB#20-008. The study was originally designed as a four-arm trial with 100 planned participants and began before COVID-19. Due to funding and safety constraints, data were collected only from exclusive smokers (n=25). Seven cases were lost due to a survey error and treated as missing at random, and we had some trials with only 24 data points for analysis. The secondary analysis protocol was approved (VT IRB#25-185).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT06910202/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT06910202/SAP_001.pdf